CLINICAL TRIAL: NCT02031757
Title: The Effectiveness of Controlled-perturbation Gait Training on Gait Rehabilitation and Fear of Falling in Individuals With Gait Impairments.
Brief Title: Effectiveness of Controlled-perturbation Gait Training on Gait Rehabilitation and Fear of Falling in Individuals With Gait Impairments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaitPert-HMO-CTIL
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2013-10

CONDITIONS: Cerebrovascular Disorders; Peripheral Nervous System Diseases; Musculoskeletal Diseases; Joint Diseases
Keywords: Balance control; Aging; Balance reactions; Perturbation
MeSH Terms: conditions — Cerebrovascular Disorders; Peripheral Nervous System Diseases; Musculoskeletal Diseases; Joint Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- perturbation training (Experimental): Standard physiotherapy augmented with perturbation training (BaMPer system).
  Interventions: Other: perturbation training
- balance exercise (Active Comparator): standard physiotherapy augmented with balance exercises.
  Interventions: Other: balance exercises

INTERVENTIONS:
Other: perturbation training — training utilizing a system that provides small, controlled and unpredictable perturbations during treadmill walking.
  Arms: perturbation training
Other: balance exercises — specific exercises regularly used in rehabilitation aiming to improve balance
  Arms: balance exercise

SUMMARY:
Gait dysfunction often occurs following stroke, neurological or musculoskeletal disease, injury and surgery. One of the consequences of such deficit is an increased risk of fall and injury. A gait training regime that incorporates controlled perturbation has been found to reduce falls in elderly population but the effectiveness of such training has yet to be studied.

The aim of this study is to evaluate the effectiveness of specific controlled dynamic perturbation training, during gait, on gait rehabilitation, fear of falling and falling with gait impaired individuals. Perturbation will be performed using a specifically designed system that provides small, controlled and unpredictable perturbations during treadmill walking.

DETAILED DESCRIPTION:
A total of 100 adults with gait dysfunction will be enrolled, evaluated and trained. They will be randomly assigned to two groups: perturbation training group and balance exercises group. Both groups will receive standard physiotherapy treatments. No gender based differences are expected so we will be able to pool male and female individuals for this analysis. Each subject of the experimental and of the control groups will be trained on 12 occasions over a period of 10-12 weeks (15 minutes, 2-3 times/week) in addition to standard care physiotherapy. Gait, balance function and fear of falling will be tested in both groups before, immediately after, 3 and 6 months after completion of the training period to explore the benefit of training.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory capability of over 2 in Functional Ambulation Classification .
* No less then 4 weeks following surgery.
* preserved mental capacity.

Exclusion Criteria:

* less then 4 weeks following surgery or injury.
* Symptomatic orthostatic hypotension, respiratory or cardiovascular, disorders that may interfere with participation in the perturbation program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
short Falls Efficacy Scale International (FES-I) | up to 6 months
  a short, easy to administer tool that measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity

SECONDARY OUTCOMES:
Berg Balance Scale | UP TO 6 MONTHS
  The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks
BalanceMaster LIMITS OF STABILITY (LOS) test | up to 6 months
  The LOS quantifies the maximum distance a person can intentionally displace their Center of Gravity without losing balance, stepping, or reaching for assistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel